CLINICAL TRIAL: NCT02415933
Title: Evaluating Child Protective Effects of Economic Strengthening and Child Rights Interventions Among Ultra-poor Families in Burkina Faso
Brief Title: Child Protective Outcomes Among Ultra-poor Families in Burkina Faso
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: TrickleUp (Unknown); Women's Refugee Commission (Unknown); Aide aux Enfants et aux Familles Démunies (ADEFAD) (Unknown); Network of European Foundations (NEF) (Unknown); Child Protection Working Group (UNICEF) (Unknown); Bernard van Leer Foundation (Unknown); Oak Foundation (Other); UBS Optimus Foundation (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB13-1481
Record Dates: First submitted 2015-03-30; First posted 2015-04-14 (Estimated); Last update posted 2024-12-31 (Actual); Status verified 2023-09

CONDITIONS: Child Abuse; Child Maltreatment
Keywords: Burkina Faso; West Africa; Children; Child Abuse; Child Mental Health; Economic Empowerment; Women's Empowerment; Domestic Violence; Child and Family Well-being; Child Separation; Child Labor; Child Maltreatment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trickle Up (Experimental): Economic empowerment
  Interventions: Behavioral: Trickle Up
- Trickle Up Plus (Experimental): Economic empowerment + child rights sensitization
  Interventions: Behavioral: Trickle Up Plus
- Wait-list (No Intervention): Women in villages assigned to the control arm do not receive any intervention during the study period, but are placed on a wait-list to receive the intervention upon completion of the evaluation phase.

INTERVENTIONS:
Behavioral: Trickle Up — Female caregivers (mothers) receive a package of interventions on economic empowerment and livelihood strengthening:
  * Savings group formation and training for a group of 15-25 women which provides a place to save, take out emergency loans and builds community networks and social capital;
  * Provision of seed grants to assist in business start-ups through microfinance loans;
  * One-on-one mentoring and coaching on livelihood development, which is held on a bi-weekly or monthly basis;
  * Trainings on financial planning and household livelihoods.
  Arms: Trickle Up
Behavioral: Trickle Up Plus — In addition to the economic empowerment program for women (Trickle Up), all members of the household assigned to Trickle Up+ arm receive sensitization component on beliefs and knowledge related to protection of children from violence and exploitation. Training sessions are developed and delivered by a local organization, Aide aux Enfants et aux Familles Démunies (ADEFAD).
  Sessions involve all members of the household and focus on knowledge and cultural norms associated with child protective outcomes (e.g. the dangers of child separation such as sending children away for work, the importance of education for girls, risks of child and forced marriage).
  Arms: Trickle Up Plus

SUMMARY:
This study tests the effects of family-based economic empowerment intervention, alone and in combination with child rights sensitization component, on child protective outcomes among ultra-poor families in Nord Region, Burkina Faso.

DETAILED DESCRIPTION:
This study evaluates a combined economic empowerment and child rights intervention to prevent violence against children and exploitation of children in ultra-poor communities in Burkina Faso. This evaluation study takes place in the Nord Region of Burkina Faso which is located in the Sahel Desert on the border to Mali. The Nord Region is characterized by extreme poverty and an ongoing food and nutrition crisis due to cyclical droughts. Extreme poverty heightens risks of violence and exploitation of children, particularly girls, who may end up in the worst forms of child labor as defined by the UN (e.g., slavery, debt bondage, forced or hazardous work in gold mines, cotton fields, or plantations in the Ivory Coast or in the South of Burkina Faso, involving physical deprivation and violence). About 1.25 million (or 37.8%) of children ages 5-14 in Burkina Faso are working to augment the incomes of their families, or because their families are too poor to support them. Adolescent girls being sent away to work as maids, facing risks of sexual exploitation and abuse. Boys being sent to religious schools madrassas, where they are made to do unpaid and/or hazardous work including begging in the street, and are subject to physical abuse.

The study employs a 3-arm cluster (group) randomized control trial design with baseline and one-year follow-up and includes 360 households (120 households per arm). Each selected household includes a female primary caregiver with a child between the ages of 10-15 who is also able to participate in the evaluation study. The study evaluates the efficacy of an economic empowerment program (Trickle Up) and a combination economic empowerment and child rights sensitization program (Trickle Up Plus) to prevent child separation and potential subsequent exposure to exploitation, abuse, and hazardous working conditions among children. Randomization occurred at the village level to assign households to three study arms: Trickle Up, Trickle Up Plus or the wait-list condition which serves as the control arm. Participants were recruited from 12 impoverished comparable villages that were selected based on socio-economic status (poverty ranking and food insecurity), geography, population size, and distance from urban center. Within these communities, families living in ultra-poverty were identified using a Participatory Wealth Ranking (PWR) exercise.

The evaluation study is implemented in partnership with the Trickle Up organization, Women's Refugee Council (WRC), and Aide aux Enfants et aux Families Démunies (ADEFAD).

ELIGIBILITY:
Inclusion Criteria:

Households that meet the following eligibility criteria will be invited to participate in the study:

1. Household meets locally defined poverty criteria (classified as an ultrapoor household);
2. Mother or female caregiver of at least one child between the ages of 10 and 15.
3. Child is between the ages of 10 and 15.
4. Male head of household provides permission for his wife and child to participate in the study;
5. Eligible child and female caregiver/parent can commit to study participation.

Exclusion Criteria:

1. Household doesn't meet locally defined poverty criteria (classified as an ultrapoor household);
2. Mother or female caregiver doesn't have at least one child between the ages of 10 and 15.
3. Child is not between the ages of 10 and 15.
4. Male head of household does not provide permission for his wife and child to participate in the study;
5. Eligible child or mother/female caregiver cannot commit to study participation.

Participants are also excluded from participation in the study if the child or the parent is assessed to have a cognitive impairment that would interfere with their ability to provide informed consent and participate in the study.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 720 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Child Protection | Baseline, 12 months, 24 months
  Questions assess children's labor-related family separation, early and forced marriage, involvement in child labor and exposure to the Worst Forms of Child Labor (e.g. slavery, debt bondage, serfdom, transactional sex, forced or hazardous work). Questions adapted from International Labour Organization (ILO)'s Statistical Information and Monitoring Programme on Child Labour (SIMPOC) Survey.
Change in Exposure to Child Abuse | Baseline, 12 months, 24 months
  Exposure to physical and emotional violence is measured using the International Society for the Prevention of Child Abuse and Neglect Screening Tool (Child Abuse Screening Tool, Children's Version / ICASTCH).

SECONDARY OUTCOMES:
Change in Child Mental Health | Baseline, 12 months, 24 months
  Child's emotional well-being and mental health problems (depression, post-traumatic symptoms and low self-esteem) are measured using Epidemiological Studies Depression Scale for Children (CES-DC), Rosenberg Self-Esteem Scale and Children's Revised Impact of Event Scale (CRIES).

OTHER OUTCOMES:
Change in Mother's Level of Depression | Baseline, 12 months, 24 months
  Change in mother's level of depression is assessed by Patient Health Questionnaire / PHQ-9
Change in Mother's Level of Anxiety | Baseline, 12 months, 24 months
  Change in mother's level of anxiety is assessed by GAD-7 Anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Ismayilova, PhD, Principal Investigator — University of Chicago
Locations (1):
- Trickle Up Burkina Faso, Ouagadougou, Burkina Faso

REFERENCES:
- [Result] Ismayilova L, Gaveras E, Blum A, To-Camier A, Nanema R. Maltreatment and Mental Health Outcomes among Ultra-Poor Children in Burkina Faso: A Latent Class Analysis. PLoS One. 2016 Oct 20;11(10):e0164790. doi: 10.1371/journal.pone.0164790. eCollection 2016. PMID 27764155
- [Result] Karimli L, Rost L, Ismayilova L. Integrating Economic Strengthening and Family Coaching to Reduce Work-Related Health Hazards Among Children of Poor Households: Burkina Faso. J Adolesc Health. 2018 Jan;62(1S):S6-S14. doi: 10.1016/j.jadohealth.2017.07.007. PMID 29273116
- [Result] Ismayilova L, Karimli L. Harsh Parenting and Violence Against Children: A Trial with Ultrapoor Families in Francophone West Africa. J Clin Child Adolesc Psychol. 2020 Jan-Feb;49(1):18-35. doi: 10.1080/15374416.2018.1485103. Epub 2018 Aug 15. PMID 30110179
- [Result] Ismayilova L, Karimli L, Sanson J, Gaveras E, Nanema R, To-Camier A, Chaffin J. Improving mental health among ultra-poor children: Two-year outcomes of a cluster-randomized trial in Burkina Faso. Soc Sci Med. 2018 Jul;208:180-189. doi: 10.1016/j.socscimed.2018.04.022. Epub 2018 May 7. PMID 29743136
- [Result] Ismayilova L, Karimli L, Gaveras E, To-Camier A, Sanson J, Chaffin J, Nanema R. An Integrated Approach to Increasing Women's Empowerment and Reducing Domestic Violence: Results of a Cluster-Randomized Controlled Trial in a West African Country. Psychol Violence. 2018 Jul;8(4):448-459. doi: 10.1037/vio0000136. Epub 2017 Aug 7. PMID 34790432
- [Result] Karimli, L., Bose, B., & Kagotho, N. (2019). Integrated Graduation Program and its Effect on Women and Household Economic Well-being: Findings from a Randomised Controlled Trial in Burkina Faso. The Journal of Development Studies, 1-18. https://doi.org/10.1080/00220388.2019.1677887
- Available data/document: Study Protocol — https://knowledge.uchicago.edu/handle/11417/69